CLINICAL TRIAL: NCT03883828
Title: Bacterial Decolonization to Prevent Radiation Dermatitis: A Randomized Controlled Trial and Quality of Life Assessment
Brief Title: Bacterial Decolonization to Prevent Radiation Dermatitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018-9722
Record Dates: First submitted 2019-02-18; First posted 2019-03-21 (Actual); Results first posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Radiation Dermatitis
MeSH Terms: conditions — Radiodermatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment Arm (Experimental): The purpose of this study is to determine whether bacterial decolonization of the nares and skin prior to treatment with radiotherapy (RT) for patients with cancers of the head and neck or breast, can prevent high-grade radiation dermatitis (RD) and improve quality of life. This study is being conducted because prior studies from this research group have found bacterial colonization in the nose prior to initiation of RT to be associated with an increased risk of high-grade RD. Patients in the treatment arm will receive pretreatment with mupirocin ointment to the nares and chlorhexidine wash to the body while patients in the control arm will receive standard of care treatment. Bacterial cultures will be taken from the nares and skin, and participants will also complete a quality of life questionnaire before and after RT.
  Interventions: Drug: Chlorhexidine gluconate solution; Drug: Mupirocin Ointment
- Control (No Intervention): Patients in the control arm will be treated according to standard of care without any radiation dermatitis prophylaxis.

INTERVENTIONS:
Drug: Chlorhexidine gluconate solution — Patients in the intervention arm will receive a decolonization regimen, consisting of intranasal mupirocin ointment to be applied twice daily to the nares and chlorhexidine wash to be used once daily to the body.
  Arms: Treatment Arm
Drug: Mupirocin Ointment — Patients in the intervention arm will receive a decolonization regimen, consisting of intranasal mupirocin ointment to be applied twice daily to the nares and chlorhexidine wash to be used once daily to the body.
  Arms: Treatment Arm

SUMMARY:
The purpose of this study is to determine whether bacterial decolonization of the nares and skin prior to treatment with radiotherapy (RT) for patients with cancers of the head and neck or breast, can prevent high-grade radiation dermatitis (RD) and improve quality of life. This study is being conducted because prior studies from this research group have found bacterial colonization in the nose prior to initiation of RT to be associated with an increased risk of high-grade RD. Patients in the treatment arm will receive pretreatment with mupirocin ointment to the nares and chlorhexidine wash to the body while patients in the control arm will receive standard of care treatment. Bacterial cultures will be taken from the nares and skin, and participants will also complete a quality of life questionnaire before and after RT.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Diagnosis of a solid tumor of the breast or head and neck with plans for fractionated radiation therapy (≥ 15 fractions) with curative intent

Exclusion Criteria:

* Prior RT to the region of interest
* Existing dermatologic condition affecting the treatment area (eg: atopic dermatitis, psoriasis, and non-healing wounds)
* Known allergy to chlorhexidine or mupirocin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2021-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth McLellan, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kost Y, Deutsch A, Mieczkowska K, Nazarian R, Muskat A, Hosgood HD, Lin J, Daily JP, Ohri N, Kabarriti R, Shinoda K, McLellan BN. Bacterial Decolonization for Prevention of Radiation Dermatitis: A Randomized Clinical Trial. JAMA Oncol. 2023 Jul 1;9(7):940-945. doi: 10.1001/jamaoncol.2023.0444. PMID 37140904

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment took place at Montefiore Medical Center between June 2019 and August 2021. The first participant was enrolled into the study on June 3, 2019
Pre-assignment Details: 80 patients were randomly assigned in a 1:1 manner to either the bacterial decolonization (treatment) arm or standard of care (control) arm. Three patients (1 assigned to the bacterial decolonization arm and 2 assigned to the control arm) were excluded from analysis because they did not start radiation therapy after enrollment. As such, the final population included 77 patients with breast cancer or head and neck cancer (39 assigned in the treatment arm and and 38 in the standard of care arm).
Groups:
- Treatment Arm: Patients in the intervention arm receive a decolonization regimen, consisting of intranasal mupirocin ointment to be applied twice daily to the nares and chlorhexidine wash to be used once daily to the body.
Period: Overall Study
Arm/Group | Treatment Arm | Control
Started | 40 | 40
Completed | 39 | 38
Not Completed | 1 | 2
Not completed — Did not start radiotherapy | 1 | 2

BASELINE CHARACTERISTICS:
Population: Baseline information and data was only collected for 77 participants (39 in the treatment arm and 38 in the control arm)
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Arm | Control | Total
Number analyzed (Participants) | 39 | 38 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.36 (10.54) | 60.42 (13.26) | 59.88 (11.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 38 | 75
  Male | 2 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 16 | 10 | 26
  Hispanic | 12 | 13 | 25
  White | 0 | 4 | 4
  Asian | 1 | 0 | 1
  Unknown | 10 | 11 | 21
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.55 (6.07) | 30.10 (5.20) | 29.45 (5.73)
Cancer Type [Count of Participants; unit: Participants]
  Breast | 38 | 37 | 75
  Head and Neck | 1 | 1 | 2
Total Radiation Dose [Median (Inter-Quartile Range); unit: Gy] | 52.4 [42.4 to 52.4] | 52.4 [42.4 to 52.4] | 52.4 [42.4 to 52.4]
Total Number of Fractions Delivered [Median (Inter-Quartile Range); unit: fractions] | 20 [16 to 20] | 20 [16 to 20] | 20 [16 to 20]
Concurrent Chemotherapy [Count of Participants; unit: Participants] | 2 | 3 | 5
Prior Chemotherapy [Count of Participants; unit: Participants] | 21 | 20 | 41
Baseline Nasal Staph. aureus Colonization [Count of Participants; unit: Participants] | 5 | 6 | 11
Silver Sulfadiazine Use [Count of Participants; unit: Participants] | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Incidence of High Grade Radiation Dermatitis
Description: The number of high-grade radiation dermatitis events (grade 2-5) were assessed at the end of treatment. Instances of Grade 2-5 radiation dermatitis was assessed using photographs taken during the final radiation therapy visit. A blinded dermatologist viewed the images and assessed for toxicity grading using CTCAE Version 5.0 criteria.
Time Frame: Last treatment session (study week depends on patient's length of treatment), approximately 5 to 8 weeks
Population: Intent to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm | Control
Number analyzed (Participants) | 39 | 38
Participants | 0 | 9
Statistical Analysis 1: Comparison: Treatment Arm vs Control; Test type: Superiority; p = 0.004, Fisher Exact — Two-sided p-values equal to or less than 0.05 were considered statistically significant; Multivariable Linear Regression = -0.45, 95% CI 2-sided [-0.75 to -0.15]

2. Primary Outcome: Median Change in Quality of Life Scoring Rated by the Skindex-16 Dermatological Survey
Description: Change in quality of life from the beginning to the end of radiation therapy was used to assess if patients receiving decolonization experienced less impact on quality of life compared to standard of care radiation therapy treatment based on the Skindex-16 survey. The Skindex-16 is a validated 16-item self-administered survey instrument that measures the effects of skin disease on patients' quality of life. Scores were determined based on changes from baseline in the three scale subcategories: Symptoms (four items, range 0-24), Emotions (seven items, range 0-42), and Functioning (five items, range 0-30) where 0 = never bothered and 6 = always bothered. Net positive changes in respective subscale scoring were correlated with an improvement in that particular Quality of life assessment (i.e., Symptoms, Emotions, Functioning), while net negative changes in scoring corresponded to a decrease in that particular Quality of life assessment.
Time Frame: From the first week (week 1) to the last week of treatment (study week depends on patient's length of treatment), approximately 5 to 8 weeks
Population: Intent to treat analysis. Data was not collected from one participant in the treatment arm and one participant in the control arm resulting in 38 and 37 participants analyzed in the treatment and control arms, respectively.
Measure: Median (Inter-Quartile Range); unit: change in score on a scale
Arm/Group | Treatment Arm | Control
Number analyzed (Participants) | 38 | 37
change in score on a scale
  Symptoms | 3 [-1 to 8] | 4 [1 to 8]
  Emotions | 5 [0 to 10] | 0 [-1 to 6]
  Functioning | 0 [0 to 2] | 0 [0 to 2]
Statistical Analysis 1: Comparison: Treatment Arm vs Control; Test type: Superiority; p = 0.20, Wilcoxon (Mann-Whitney) — A 2-sided P ≤ .05 was considered statistically significant; Symptoms Domain
Statistical Analysis 2: Comparison: Treatment Arm vs Control; Test type: Superiority; p = 0.05, Wilcoxon (Mann-Whitney) — A 2-sided P ≤ .05 was considered statistically significant; Emotions Domain
Statistical Analysis 3: Comparison: Treatment Arm vs Control; Test type: Superiority; p = 0.73, Wilcoxon (Mann-Whitney) — A 2-sided P ≤ .05 was considered statistically significant; Functioning Domain

ADVERSE EVENTS:
Time Frame: The adverse event monitoring period spanned the duration of the intervention (5 days before radiotherapy start and until the last day of radiotherapy) for each patient. This varies per patient between 5 to 8 weeks.
Arm/Group | Treatment Arm | Control
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/38
Other Adverse Events (participants affected / at risk) | 1/39 | 0/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=39) | Control (N=38)
Itch (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-13): https://cdn.clinicaltrials.gov/large-docs/28/NCT03883828/Prot_SAP_000.pdf